CLINICAL TRIAL: NCT00957736
Title: Targeted Single Nucleotide Polymorphisms (SNPs) to Classify Subtypes of Chronic Graft-Versus-Host Disease (cGVHD) After Allogeneic Transplant.
Brief Title: Chronic Graft-Versus-Host Disease in Patients Who Have Undergone Donor Stem Cell Transplant
Status: Terminated | Type: Observational
Why Stopped: study closed prematurely upon PI's departure from VICC
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Madan Jagasia, MD, Associate Professor of Medicine, Medical Oncologist, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC BMT 0867; P30CA068485 (NIH); VU-VICC-BMT-0867; IRB# 080995
Record Dates: First submitted 2009-08-11; First posted 2009-08-12 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Cancer
Keywords: graft versus host disease; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Hodgkin lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; recurrent/refractory childhood Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; noncontiguous (NC) stage II adult Burkitt lymphoma; NC stage II adult diffuse large cell lymphoma; NC stage II adult diffuse mixed cell lymphoma; NC stage II adult diffuse small cleaved cell lymphoma; NC stage II adult immunoblastic large cell lymphoma; NC stage II adult lymphoblastic lymphoma; NC stage II grade 1 follicular lymphoma; NC stage II grade 2 follicular lymphoma; NC stage II grade 3 follicular lymphoma; NC stage II mantle cell lymphoma; NC stage II marginal zone lymphoma; NC stage II small lymphocytic lymphoma; accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); atypical chronic myeloid leukemia, BCR-ABL negative; blastic phase chronic myelogenous leukemia; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; juvenile myelomonocytic leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; childhood myelodysplastic syndromes; chronic eosinophilic leukemia; primary myelofibrosis; chronic neutrophilic leukemia; de novo myelodysplastic syndromes; disseminated neuroblastoma; myelodysplastic/myeloproliferative neoplasm, unclassifiable; poor prognosis metastatic gestational trophoblastic tumor; previously treated childhood rhabdomyosarcoma; previously treated myelodysplastic syndromes; recurrent Wilms tumor and other childhood kidney tumors; recurrent childhood rhabdomyosarcoma; recurrent neuroblastoma; recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; recurrent malignant testicular germ cell tumor; secondary myelodysplastic syndromes; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; stage III malignant testicular germ cell tumor; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; refractory multiple myeloma
MeSH Terms: conditions — Neoplasms; Graft vs Host Disease; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Recurrence; Mycosis Fungoides; Sezary Syndrome; Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelomonocytic, Juvenile; Leukemia, Myeloid, Acute; Leukemia, Hairy Cell; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Neutrophilic, Chronic; Myeloproliferative Disorders; Wilms Tumor; Neuroblastoma; Carcinoma, Ovarian Epithelial; Testicular Neoplasms; Multiple Myeloma; Breast Neoplasms | interventions — Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Allogeneic stem cell transplant: Stem cells from a genetically non-identical donor transplanted into a patient.
  Interventions: Genetic: polymorphism analysis; Other: laboratory biomarker analysis

INTERVENTIONS:
Genetic: polymorphism analysis — Will assess the SNPs present in both the donor and to host and correlate the SNPs with outcome based in the NIH consensus criteria for cGVHD. Candidate SNPs will include but are not limited to TGF-β18, mannose binding lectin19, myeloperoxidase, HSP 70, minor histocompatability antigens, KIR, CCL513, NOD2/CARD1512, TNFα11, TNF R II, IL-1010, 11, IL-1317, IL-620, IFN-γ20, IL-1 RA21, IL-2315, and IL-1516. Other candidate genes will be assessed on current review of the literature and candidate SNPs will be added based on their relationship to aGVHD, cGVHD, autoimmune disease, pharmacogenetics, and other immunologic processes. The genes will be assessed for gene frequency using the HapMap and SNP databases prior to statistical analysis.
Other: laboratory biomarker analysis — Will assess the SNPs present in both the donor and to host and correlate the SNPs with outcome based in the NIH consensus criteria for cGVHD. Candidate SNPs will include but are not limited to TGF-β18, mannose binding lectin19, myeloperoxidase, HSP 70, minor histocompatability antigens, KIR, CCL513, NOD2/CARD1512, TNFα11, TNF R II, IL-1010, 11, IL-1317, IL-620, IFN-γ20, IL-1 RA21, IL-2315, and IL-1516. Other candidate genes will be assessed on current review of the literature and candidate SNPs will be added based on their relationship to aGVHD, cGVHD, autoimmune disease, pharmacogenetics, and other immunologic processes. The genes will be assessed for gene frequency using the HapMap and SNP databases prior to statistical analysis.

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to chronic graft-versus-host disease in patients who have undergone donor stem cell transplant.

PURPOSE: This phase I trial is studying chronic graft-versus-host disease in patients who have undergone donor stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine and define the biological basis of different subtypes of chronic graft-vs-host disease using a targeted single nucleotide polymorphisms approach in patients who have undergone allogeneic stem cell transplantation.

OUTLINE: Two important aspects of the methodologies that will be employed for the analysis of SNPs associated with GVHD are throughput efficiency to be able to perform the assays on a reasonable number of samples as well as having the ability to add or remove SNPs to the assay panel. While a genome-wide association study to identify variants associated with GVHD would offer an unbiased approach, our patient cohort size would not allow significant statistical power in the study. Therefore, a more targeted approach using two established technologies is proposed.

The Sequenome assay uses the unique combination of a single-base primer extension assay incorporating one of four modified nucleotides. The four modified nucleotides each have a unique mass that allows them to be distinguished from one another using mass spectrometry. Each SNP is determined analyzing the primer extension product from a PCR amplicon that surrounds the SNP of interest. The development of each assay involves designing flanking PCR primers and an internal extension assay using web-based software provided by Sequenome. The assays can be designed to analyze up to 30 SNPs in a single reaction, providing a customizable, efficient and high-throughput assay for SNPs of interest.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Underwent prior matched related or unrelated allogeneic stem cell transplantation (SCT)

  * Presence OR absence of chronic graft-vs-host disease after day 100 and alive after day 180 post-transplantation
* No T-cell depleted SCT, cord blood transplantation, mismatched allogeneic transplantation, or autologous transplantation
* Available recipient and donor DNA (samples collected from the Vanderbilt University or the Fred Hutchinson Cancer Center tissue bank)

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: allogeneic stem cell transplant patients
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2008-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To study the SNP profiles of a select group of candidate non-HLA genes among various cGVHD subtypes. Patients will be stratified as having classic cGVHD vs. non-classic GVHD for initial analyses. | Upon data collection of final patient

SECONDARY OUTCOMES:
Correlation of SNP profiles with predominant organ involvement and responsiveness of cGVHD to therapy | Upon collection of data on final patient
Correlation of SNP profiles with survival endpoints | Upon collection of data on final patient

CONTACTS AND LOCATIONS:
Overall Officials: Madan Jagasia, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee